CLINICAL TRIAL: NCT05420285
Title: Cardiometabolic Effects of Dapagliflozin in Heart Failure With Reduced or Mildly Reduced Ejection Fraction: an Exploratory Study
Brief Title: Cardiometabolic Effects of Dapagliflozin in Heart Failure With Reduced or Mildly Reduced Ejection Fraction
Acronym: ICARD
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: APHP210166; 2021-000481-14 (EudraCT Number)
Record Dates: First submitted 2022-05-12; First posted 2022-06-15 (Actual); Last update posted 2022-12-09 (Actual); Status verified 2022-02

CONDITIONS: Heart Failure; Reduced Ejection Fraction
Keywords: heart failure; HFrEF; myocardial function; fibrosis; metabolism
MeSH Terms: conditions — Heart Failure; Fibrosis | interventions — dapagliflozin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dapagliflozin (Experimental): Dapagliflozin is taken orally, once daily at the dosage of 10 mg during 6 months.
  Interventions: Drug: Dapagliflozin

INTERVENTIONS:
Drug: Dapagliflozin — Dapagliflozin (Forxiga) is a very potent selective and reversible inhibitor of SGLT2.
  Other Names: Forxiga

SUMMARY:
Gliflozins have demonstrated a beneficial effect in terms of incident heart failure and related events in patients with or without diabetes. The clinical trial ICARD is an exploratory study that aims to evaluate the cardiometabolic mechanistic effects on the myocardium of dapagliflozin in heart failure with reduced ejection fraction. Deep phenotyping of cardiac and vascular function will be performed using MRI. Myocardial tissue characterization will be based on MRI and FDG-PET for glucose metabolism assessment. Liver steatosis and fibrosis will simultaneously be assessed.

DETAILED DESCRIPTION:
Open-label, non-controlled clinical trial (Jardé 1) to assess the cardiovascular and metabolic effects of once-daily dapagliflozin 10 mg during 6 months in patients with heart failure and reduced ejection fraction.

Eligibility of patients addressed to the Department of Cardiology (Prof R. Isnard, Pitié-Salpêtrière Hospital, Paris, France) will be investigated at V0: inclusion and exclusion criteria will be checked and informed consent will be signed.

Up to twenty one days after V0, patients will come to the VMRI visit (VMRI) for the cardiac and liver gadolinium-injected MRI and AGE Reader (VRMI) and to the baseline visit (V1). Pregnancy will be ruled out in women of childbearing potential with blood beta-HCG. A blood test (including metabolomics and lipidomics) and FDG-PET MRI including Glucose Tolerance Test (GTT) will be performed. Dapagliflozin 10 mg once daily during six months will be prescribed.

Fifteen to twenty-one days after treatment initiation, a safety visit (V2) will take place in order to verify the tolerance.

A pre-final visit (V3) will be organized after a total of 23 weeks (± 1 week) of treatment. Pregnancy will be ruled out in women of childbearing potential with blood beta-HCG. A blood test (including metabolomics and lipidomics), ECG, trans-thoracic echocardiography (TTE), cardiac and liver MRI and AGE Reader will be performed.

After 24 weeks of treatment (6-month treatment), patients will come to the end of study visit (V4), to undergo the final FDG-PET MRI including Glucose Tolerance Test (GTT).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* NYHA functional class II-IV.
* Previous hospitalization for heart failure anytime or NT-proBNP >125 pg/ml in the previous 12 months
* Left ventricular ejection fraction ≤ 50% measured at least 1 time in transthoracic echocardiography in the last 12 months
* Treated by optimal medical therapy (ACE-I or angiotensin receptor blocker or sacubitril-valsartan, and betablockers, and mineralocorticoid receptor antagonist and furosemide) unless such use was contraindicated or previously associated with side-effects leading to drug discontinuation. No change in drugs dosages in the last month.
* Able to give written informed consent
* If female of childbearing potential, have a negative serum pregnancy test
* Use of a validated method of birth control until the end of the study (men and women)
* Affiliation to a social security regime

Exclusion Criteria:

* Hypersensitivity to dapagliflozin or to any of the excipients
* Current treatment with gliflozine
* Cardiac rhythm disorder including atrial fibrillation > 100 bpm
* Significant valvular heart disease including mitral or aortic regurgitation > II/IV
* Hospitalisation for heart failure or unplanned visit for worsening heart failure in the last month
* Recent (last 3 months) or planned coronary revascularization
* Acute coronary syndrome, stroke, or transient ischemic attack in the last 3 months
* Body mass-index > 40 kg/m2
* Uncontrolled type 2 diabetes (Hb1AC > 9%) or type 1 diabetes
* Genetic diabetes (Maturity Onset Diabetes of the Young, MODY)
* Current treatment for cancer, cardiotoxic cancer treatment in the last year
* Treatment with systemic steroids at time of informed consent or change in dosage of thyroid hormones in the last 6 weeks
* Active infectious diseases
* Hypovolemia or dehydration, severe hypokalaemia, or severe hyponatremia
* Contraindication to MRI or to contrast agents used
* Estimated glomerular filtration rate (eGFR) < 30 ml per minute per 1.73 m2 of body-surface area (according to the Modification of Diet in Renal Disease criteria)
* Patient on AME (state medical aid)
* Pregnant or breast-feeding female
* Current participation in another interventional study or being in the exclusion period at the end of a previous study
* Patient protected by law (guardianship, tutelage measure, deprived of liberty)

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-06-26 (Actual); Primary Completion 2023-09 (Estimated); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
To evaluate changes in left ventricular (LV) extracellular mass index (ECMi) measured by MRI, induced by once-daily dapagliflozin 10mg during 6 months in patients with heart failure and reduced ejection fraction | 6 months
  MRI measurement of changes in left ventricular extracellular mass index (ECMI) after a 6-month once-daily dapagliflozin 10 mg regimen

SECONDARY OUTCOMES:
To evaluate myocardial morphology | 6 months
  MRI measurement of change: Left and right ventricular volumes and Left atrial volumes
To evaluate myocardial morphology | 6 months
  MRI measurement of change: LV mass
Left ventricular ejection fraction as a biomarker of myocardial function | 6 months
  MRI measurement of change of left ventricular ejection fraction
Right ventricular ejection fraction as a biomarker of myocardial function | 6 months
  MRI measurement of change of right ventricular ejection fraction
Left atrial ejection fraction as a biomarker of myocardial function | 6 months
  MRI measurement of change of left atrial ejection fraction
Peak global longitudinal strain as a biomarker of myocardial function | 6 months
  MRI measurement of change of peak global LV longitudinal strain
Peak radial strain as a biomarker of myocardial function | 6 months
  MRI measurement of change of peak radial LV strain
Peak circumferential strain as a biomarker of myocardial function | 6 months
  MRI measurement of change of peak circumferential LV strain
Peak circumferential strain as a biomarker of left atrial function | 6 months
  MRI measurement of change of peak circumferential LA strain (reservoir)
Peak circumferential strain as a biomarker of left atrial function | 6 months
  MRI measurement of change of peak circumferential LA strain (booster)
LV myocardial dense fibrosis (late gadolinium enhancement) as a biomarker of fibrosis | 6 months
  MRI measurement of change of LV myocardial dense fibrosis (late gadolinium enhancement mass)
Intracellular mass index (ICMi) as a biomarker of fibrosis | 6 months
  MRI measurement of change of intracellular mass index (ICMi)
Extracellular mass index (ECMi) as a biomarker of fibrosis | 6 months
  MRI measurement of change of extracellular mass index (ECMi)
To evaluate adipose tissue | 6 months
  MRI measurement of change: epicardial adipose tissue (EAT) and steatosis (triglyceride fraction)
To evaluate myocardial steatosis | 6 months
  1H-MR spectromscopy measurement of modifications of relative myocardial triglyceride content.
To evaluate glucose metabolism | 6 months
  18FDG-PET-MRI measurement of change with glucose uptake analysis
Effects of dapagliflozin therapy on the proximal aorta | 6 months
  High resolution cine aortic MRI measurement of ascending aortic areas
Effects of dapagliflozin therapy on the proximal aorta | 6 months
  High resolution cine aortic MRI measurement of descending aortic areas
Effects of dapagliflozin therapy on the proximal aorta | 6 months
  High resolution cine aortic MRI measurement of ascending aortic distensibility
Effects of dapagliflozin therapy on the proximal aorta | 6 months
  High resolution cine aortic MRI measurement of descending aortic distensibility
Effects of dapagliflozin therapy on the proximal aorta | 6 months
  High resolution cine aortic MRI measurement of aortic arch pulse wave velocity (PWV)
To evaluate the evolution of body composition in multimodality imaging | 6 months
  MRI measurement of change in abdominal subcutaneous and visceral fat using the ATQUA method on DIXON MRI images
To evaluate the changes in fasting glucagon | 6 months
  Blood measurement change in glucagon
To evaluate the changes in fasting β-hydroxybutyrate | 6 months
  Blood measurement change in β-hydroxybutyrate
To evaluate the changes in fasting glycerol | 6 months
  Blood measurement change in glycerol
To evaluate the changes in free fatty acid (FFA) | 6 months
  Blood measurement change in free fatty acid (FFA)
To evaluate the changes in fasting glycemia | 6 months
  Blood measurement change in glycemia
To evaluate the subcutaneous tissue Advanced end-Glycation Products (AGE) | 6 months
  Measurement of the value of AGE on AGE reader
Evaluation of pathophysiological changes at the molecular level (metabolite profiling) | 6 months
  Blood measurement of targeted metabolites by LC-MS (Liquid chromatography coupled to mass spectrometry) and by GC-MS (Gas chromatography coupled to mass spectrometry)

CONTACTS AND LOCATIONS:
Overall Officials: Alban REDHEUIL, MD PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Pitié-Salpêtrière Hospital, Paris, France

IPD SHARING:
Plan to Share IPD: Yes
Data are available upon reasonable request. The procedures carried out with the French data privacy authority (CNIL, Commission Nationale de l'Informatique et des Libertés) do not provide for the transmission of the database, nor do the information and consent documents signed by the patients.
  Consultation by the editorial board or interested researchers of individual participant data that underlie the results reported in the article after deidentification may nevertheless be considered, subject to prior determination of the terms and conditions of such consultation and in respect for compliance with the applicable regulations.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Beginning 3 months and ending 3 years following article publication. Requests out of these time frame can also be submitted to the sponsor
Access Criteria: Researchers who provide a methodologically sound proposal